CLINICAL TRIAL: NCT00005329
Title: Protein S and Myocardial Infarction
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4128; R01HL030443 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2005-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Myocardial Infarction
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Myocardial Infarction

SUMMARY:
To test the hypothesis that low levels of free protein S, a natural anticoagulant protein in plasma, were associated with an increased incidence of myocardial infarction in middle aged men and women.

DETAILED DESCRIPTION:
BACKGROUND:

Free protein S (that portion of plasma protein S which is not in complex with C4b binding protein) is a cofactor for the anticoagulant effect of activated protein C. Patients presenting with acute myocardial infarction have significantly reduced levels of free protein S. If the major hypothesis proved correct, patients at high risk of myocardial infarction could be identified and could be targeted for future studies to examine specific intervention therapy.

DESIGN NARRATIVE:

The blinded and prospective study began in 1992, although the grant was first awarded in 1983. The goal was to determine if low levels of free protein S were associated with an increased incidence of myocardial infarction. Plasma samples were obtained yearly from 2,224 men aged 50-59 years who were participants in the Second Northwick Park Heart Study sponsored by the British Medical Research Council Epidemiology and Medical Care Unit. Clinical endpoints for the study were documented fatal and non-fatal myocardial infarction. To prevent potential bias, this laboratory was blinded to the clinical endpoints until all samples had been collected and all causes of death in the study population had been adjudicated. ln addition to free protein S, total protein S and C4b binding protein were measured. The study design permitted the assessment of the temporal relationship between the development of low free protein S levels and the occurrence of myocardial infarction and the presence or absence of a biologic gradient (dose-response) between levels of free protein S and the frequency of infarction. These two analyses were important in assessing whether the observed association was causal or whether low protein S occured as a consequence of myocardial infarction. Three levels of free protein S had been defined prior to initiating the study to determine if the frequency of myocardial infarction did follow a biologic gradient. The measurement of other potential markers of risk by other laboratories, such as prothrombin fragment Fl+2 and factor X activation peptide, permitted a comprehensive evaluation of hemostatic risk factors in myocardial infarction. A second study was conducted in women to examine protein S as a risk factor for myocardial infarction.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1992-05; Study Completion 1997-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Comp — University of Oklahoma Hlth Sciences Ctr

REFERENCES:
- [Background] Eichner JE, Moore WE, McKee PA, Schechter E, Reynolds DW, Qi H, Comp PC. Fibrinogen levels in women having coronary angiography. Am J Cardiol. 1996 Jul 1;78(1):15-8. doi: 10.1016/s0002-9149(96)00219-6. PMID 8712111
- [Background] Thorisdottir H, Evans JA, Schwartz HJ, Comp P, Haluschak J, Ratnoff OD. Some clotting factors in plasma during danazol therapy: free and total protein S, but not C4b-binding protein, are elevated by danazol therapy. J Lab Clin Med. 1992 Jun;119(6):698-701. PMID 1534346
- [Background] Rudnicka AR, Miller GJ, Nelson T, Doray D, Comp PC. An association between plasma free protein s concentration and risk of coronary heart disease in middle-aged men. Thromb Res. 2001 Jan 15;101(2):1-11. doi: 10.1016/s0049-3848(00)00379-0. PMID 11342201